CLINICAL TRIAL: NCT02614937
Title: Open Label Squalamine Lactate Ophthalmic Solution for the Treatment of Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO) and Central Retinal Vein Occlusion (CRVO)
Brief Title: Study of Squalamine Lactate for the Treatment of Macular Edema Related to Retinal Vein Occlusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohr Pharmaceutical Inc. (Industry)
Collaborators: Cumberland Valley Retina Consultants, PC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHR-004
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Squalamine and ranibizumab to Week 10 (Experimental): All eyes received an initial 10 week mandatory loading period of topical Squalamine Lactate Ophthalmic Solution, 0.2% therapy.
  All eyes received mandatory intravitreal injections of ranibizumab 0.5mg at the conclusions of weeks 2 and 6.
  Randomize at Week 10 to 2 different groups - Squalamine and No Squalamine, continue PRN ranibizumab in both groups
  Interventions: Drug: ranibizumab; Drug: Squalamine Lactate Ophthalmic Solution, 0.2%
- Continue Squalamine, ranibizumab PRN (Experimental): Continue use of Squalamine Lactate Ophthalmic Solution, 0.2% after Week 10; continue ranibizumab 0.5 mg IVT PRN
  Interventions: Drug: ranibizumab
- Stop Squalamine, ranibizumab PRN (Experimental): Discontinue use of Squalamine Lactate Ophthalmic Solution, 0.2% after Week 10; continue ranibizumab 0.5 mg IVT PRN
  Interventions: Drug: ranibizumab; Drug: Squalamine Lactate Ophthalmic Solution, 0.2%

INTERVENTIONS:
Drug: ranibizumab — 0.5 mg IVT ranibizumab
  Other Names: Lucentis
Drug: Squalamine Lactate Ophthalmic Solution, 0.2% — Squalamine Lactate Ophthalmic Solution BID
  Arms: Squalamine and ranibizumab to Week 10; Stop Squalamine, ranibizumab PRN

SUMMARY:
This was a prospective, single center, open label, randomized study evaluating the biological effect of squalamine lactate ophthalmic solution, 0.2% combined with intravitreous ranibizumab in patients with macular edema secondary to branch, hemi-central and central retinal vein occlusion (BRVO, HRVO, CRVO).

DETAILED DESCRIPTION:
At baseline, all eyes underwent ETDRS visual acuity measurements at 4 meters, a complete ophthalmological evaluation, SD-OCT imaging of the macula, and fluorescein angiographic assessment of capillary perfusion in the macula and peripheral fundus. All eyes received an initial 10 week mandatory loading period of topical squalamine therapy.

All eyes received mandatory intravitreal injections of ranibizumab 0.5mg at the conclusions of weeks 2 and 6. At the conclusion of week 10, eyes were randomized in a 1:1 ratio to continue squalamine drops bid or discontinue squalamine drops in the study eye. All eyes were examined every 4 weeks through the week 38 endpoint and were eligible to receive additional as needed ranibizumab 0.5mg injections starting at the conclusion of week 10 and every 4 weeks thereafter through week 34 depending upon prespecified visual acuity and OCT retreatment criteria.

Any eye with a decrease of 5 or more ETDRS letters or increase in CST on OCT of 50uM or more from their best previous measurements automatically received an additional ranibizumab 0.5mg injection beginning at the conclusion of week 10.

Eyes randomized to continue squalamine drops did so through the week 38 endpoint. SD-OCT measurements of the macula were obtained at every study visit. Fluorescein angiograms were performed on the study eye at baseline, weeks 10 and 38.

Safety endpoints included all adverse events spontaneously reported, elicited or observed were documented by the investigators at any visit.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with treatment naïve, center involving macular edema secondary to BRVO, HRVO or CRVO in patients of at least 40 years of age
* Macular edema of 1-4 months duration prior to the baseline visit
* Best corrected baseline ETDRS visual acuity of 20/40 to 20/320 Snellen equivalent using the 4 meter testing method
* Baseline CST greater than or equal to 325uM using SD-OCT imaging
* Less than 50% foveal capillary ring disruption as defined by fluorescein angiography (FA)
* Absence of dense intraretinal or subretinal hemorrhage and or lipid through the foveal center
* Absence of subfoveal fibrosis or hyperpigmentation.

Exclusion Criteria:

* Eyes with ocular pathology other than RVO related macular edema such as clinically significant cataract or media opacity, diabetic retinopathy, macular degeneration, glaucoma, uveitis, epiretinal membrane, vitreomacular traction or intraocular tumor
* Intraocular surgery within 6 months prior to baseline
* Two-plus or greater afferent pupillary defect (APD) in the study eye
* Likelihood of evidence driven indication for peripheral scatter photocoagulation within 6 months of recruitment
* History of previous intravitreal pharmacologic treatment of any kind in the study eye
* History of previous retinal laser photocoagulation of any kind in the study eye
* History of intravitreal anti-VEGF therapy in the fellow eye within 6 months prior to baseline
* Any evidence of baseline ocular neovascularization such as disc neovascularization, preretinal neovascularization, iris or angle neovascularization in the study eye
* Eyes that have shown spontaneous improvement within the preceding 3 months defined as an improvement of best corrected visual acuity of greater than 15 ETDRS letters or thinning of the CST on OCT of greater than 20%

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Visual Function - Efficacy | Baseline to Week 38
  Mean change in ETDRS letter score from baseline

SECONDARY OUTCOMES:
Visual Function - Efficacy | Baseline to Week 38
  Eyes with visual outcomes of 20/40 or better at Week 38 compared to Baseline Visit
Retinal Anatomy - Efficacy | Baseline to Week 38
  Proportion of eyes with Central Subfield Thickness (CST) on SD-OCT less than 325 microns at Week 38
Safety and Tolerability as measured by adverse event reporting and ophthalmologic examination from Baseline to Week 38 | Baseline to Week 38
  Safety as measured by adverse event reporting and ophthalmologic examination from Baseline to Week 38
Concomitant ranibizumab administration - efficacy | Baseline to Week 38
  Number of injections of 0.5 mg ranibizumab to keep edema resolved from Week 2 through Week 34 of study

CONTACTS AND LOCATIONS:
Overall Officials: John Wroblewski, MD, Principal Investigator — Cumberland Valley Retinal Consultants, Hagerstown, MD